CLINICAL TRIAL: NCT01636882
Title: A Phase 2 Study of the Efficacy and Safety of Intratumoral CAVATAK™ (Coxsackievirus A21, CVA21) in Patients With Stage IIIc and Stage IV Malignant Melanoma to Extend Dosing for up to 48 Weeks Total (VLA-008 CALM Ext)
Brief Title: CAVATAK in Patients With Stage IIIc or IV Malignant Melanoma to Extend Dosing to 48 Weeks (VLA-008 CALM Ext)
Acronym: CALMext
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-006-Ext; VLA-008 (Other: Viralytics Study ID)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Melanoma
Keywords: Melanoma; CALM
MeSH Terms: conditions — Melanoma

ARMS (1):
- CVA21 (Experimental): Dose of CAVATAK up to 3 x 10⁸ TCID50 for an additional 9 treatments at 3-week intervals
  Interventions: Biological: CVA21

INTERVENTIONS:
Biological: CVA21

SUMMARY:
This is an extended use study for patients who have received 10 doses of CAVATAK™ in the VLA 007 trial. There may be patients who have benefitted from the study drug and who might benefit from further treatment. In order to accommodate those patients further treatment to complete 48 weeks of CVA21 intratumoral injections will be made available.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have reached Week 24 of the core protocol in immune-related complete response (irCR), immune-related partial response (irPR), immune-related stable disease (irSD), or immune-related progressive disease (irPD) (unconfirmed) with evidence of tumor inflammatory reaction.
* 2. If patient is in irPD (unconfirmed) status, they must not have had a decrease in their Karnofsky Performances Scale (KPS) score > 10 points and to be judged to not have "rapid clinical deterioration" by the investigator since the subject's last tumor measurement leading to irPD assessment.
* 3. Patients must start treatment in the extension protocol within 8 weeks of their last injection administered in the core protocol.
* 4. Patient is able and willing to provide written informed consent to participate in the study.
* 5. Fertile males and females must agree to the use of an adequate form of contraception, e.g., condoms for males.

Exclusion Criteria:

* 1. Tumors to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigators, could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis.
* 2. If lesions are too small to be visualized or palpable for accurate injection.
* 3. Currently in status of irPD (confirmed) or irPD (unconfirmed) without evidence of tumor inflammatory response, or with rapid clinical deterioration, or with a decrease of 10 points or more on their KPS score since their last assessment before irPD (unconfirmed) assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07-03 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Oncology Specialists, Park Ridge, Illinois
  - Providence Medical Centre, Portland, Oregon
  - Mary Crowley Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Andtbacka RHI, Curti B, Daniels GA, Hallmeyer S, Whitman ED, Lutzky J, Spitler LE, Zhou K, Bommareddy PK, Grose M, Wang M, Wu C, Kaufman HL. Clinical Responses of Oncolytic Coxsackievirus A21 (V937) in Patients With Unresectable Melanoma. J Clin Oncol. 2021 Dec 1;39(34):3829-3838. doi: 10.1200/JCO.20.03246. Epub 2021 Aug 31. PMID 34464163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical clinics from 03 July 2012 to 29 July 2015 (last subject enrolled in VLA-008).
Pre-assignment Details: Subjects were screened for and excluded from the study if they had pre-existing antibodies to CVA21.
Groups:
- CVA21: Dose of CVA21 up to 3 x 10⁸ TCID50 for an additional 9 treatments at 3-week intervals
Period: Overall Study
Arm/Group | CVA21
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CVA21: Dose of CAVATAK up to 3 x 10⁸ TCID50 for an additional 9 treatments at 3-week intervals CVA21
Arm/Group | CVA21
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Participants with Grade 3 or Higher Adverse Events
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | CVA21
Number analyzed (Participants) | 16
participants | 16

ADVERSE EVENTS:
Time Frame: 1 year
Description: Listed serious adverse events (SAEs) and adverse events (AEs) are irrespective of treatment relationship. No SAEs reported were attributable to CVA21. No serious unexpected adverse events (SUSARs) were reported for the study.
Arm/Group | CVA21
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=16)
Cardiac arrest (Cardiac disorders) | 1 (1)
Motor Dysfunction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=16)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Chills (General disorders) | 2 (4)
Influenza like illness (General disorders) | 2 (3)
Chest discomfort (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (2)
Injection site inflammation (General disorders) | 1 (1)
Injection site oedema (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (6)
Injection site pruritus (General disorders) | 1 (1)
Injection site vesicles (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Motor dysfunction (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Occult blood (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes